CLINICAL TRIAL: NCT05883306
Title: A Clinical Trial to Assess Absorption, Metabolism and Excretion of [14C]-LXI-15028 in Chinese Healthy Male Subjects - Mass Balance and Biotransformation Study of [14C]LXI-15028 in Humans
Brief Title: Mass Balance and Biotransformation Study of [14C]LXI-15028 in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Luoxin Pharmaceutical Group Stock Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NE822201
Record Dates: First submitted 2023-05-10; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Healthy Subjects; Pharmacokinetics of 14C-labeled of LXI-15028

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]LXI-15028(n=6-8) (Experimental): Subjects will receive a single oral dose of [14C]LXI-15028 suspension under the fasted state .
  Interventions: Drug: [14C]LXI-15028

INTERVENTIONS:
Drug: [14C]LXI-15028 — [14C]LXI-15028

SUMMARY:
To assess absorption, metabolism and excretion of [14C]-LXI-15028 in Chinese healthy male Subjects following a single oral dose of [14C]LXI-15028 suspension.

ELIGIBILITY:
Inclusion Criteria:

* Chinese healthy male subjects;
* 18 to 45 years of age (inclusive)
* Body mass index (BMI) of 19-26 kg/m2 (inclusive), and body weight not less than 50 kg (inclusive)
* Voluntarily signing the ICF
* Ability to communicate well with the investigator and compliance to complete the trial according to the protocol.

Exclusion Criteria:

* Clinically significant abnormality of physical examination, vital signs, routine laboratory tests (hematology, blood chemistry, coagulation, urinalysis, stool routine + occult blood, and thyroid function), 12-lead ECG, chest CT, and abdomen ultrasound (liver, gallbladder, pancreas, spleen, and kidneys), etc.
* Resting QT interval (QTcF) ≥ 450 ms by 12-lead electrocardiogram (ECG)
* Hepatitis B surface antigen or hepatitis B e antigen test, hepatitis C virus antibody IgG test, human immunodeficiency virus antigen/antibody combination test, or Treponema pallidum antibody test is positive
* Novel coronavirus infection screening shows C-reactive protein is clinically significant abnormality, or COVID-19 nucleic acid test is positive
* Use of any drugs inhibiting or inducing hepatic drug metabolizing enzymes within 30 days before screening;
* Use of any prescription drugs, over-the-counter drugs, Chinese herbal medicines, or dietary supplements such as vitamins and calcium supplements within 14 days before screening;
* History of any clinical critical illness or presence of diseases or conditions that the investigator considers may affect the trial results, including but not limited to diseases of cardiovascular system, circulatory system, respiratory system, endocrine system, nervous system, digestive system, urinary system or blood, immune system, and psychiatric system, especially metabolism and nutrition diseases and gastrointestinal diseases;
* Major surgery within 6 months before screening or incomplete healing of surgical incision, the major surgeries including but not limited to any procedures that have significant risk of hemorrhage, prolonged general anesthesia, open biopsy, or marked traumatic invasive injury;
* Subjects with an allergic constitution (e.g., history of bronchial asthma, allergy to food and pollen, allergy to two or more drugs, or history of allergy), including any previous serious adverse reaction to proton pump inhibitors or potassium-competitive acid blockers (e.g., omeprazole, rabeprazole, lansoprazole, and vonoprazan), or known hypersensitivity to penicillin or cephalosporin antibiotics; or those who may be hypersensitive to the investigational drug or its excipients, as judged by the investigator;
* Hemorrhoids or perianal diseases with regular/current hematochezia, irritable bowel syndrome, and inflammatory bowel disease;
* Habitual constipation or diarrhea;
* Alcoholism or frequent alcohol use within 6 months before screening, i.e., weekly alcohol consumption > 14 units (1 unit = 360 mL of beer or 45 mL of ABV 40% spirit or 150 mL of wine); or positive alcohol breath test result at Screening;
* Daily smoking exceeding 5 cigarettes (≥ 5 cigarettes) within 3 months before Screening, or habitual use of nicotine-containing products and inability to withdraw during the trial period;
* Drug abuse, use of soft drug (e.g., marijuana) within 3 months before screening, or use of hard drug (e.g., cocaine, amphetamines, phencyclidine, etc.) within 1 year before screening; or positive urine drug test at screening;
* Drinking excessive tea, coffee and/or caffeine-containing beverages (over 8 cups, 1 cup = 250 mL) on a daily basis within 3 months prior to screening;
* Inability to avoid intake of grapefruit, bitter orange, starfruit, pithya, mango, and other fruit or fruit juice that may affect the metabolism from 7 days before administration until completion of the study;
* Work with long-term exposure to radioactive conditions; or marked exposure to radioactivity (chest/abdomen CT ≥ 2 times, or other kinds of X-ray examinations ≥ 3 times) or participation in any radioactive labeling trial within 1 year before the trial;
* History of fear of needles and blood, difficult blood sampling, or incapability of tolerating blood sampling via venipuncture;
* Participation in any other clinical trial (including drug and device clinical trials) within 3 months before screening;
* Vaccination within 1 month before Screening or planned vaccination during the trial period;
* Subjects who have a plan for parenthood or sperm donation from the signing of informed consent to 1 year following the completion of the trial, or those who do not agree that subjects and their partners should use strict contraception from the signing of informed consent to 1 year following the completion of the trial;
* Blood loss or blood donation up to 400 mL (≥ 400 mL) within 3 months before Screening, or blood transfusion within 1 month before screening;
* Subjects who have any factors that make them not suitable for participating in this trial, as assessed by the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Mass balance | approximately 11 days
  Mass balance recovery of total radioactivity in urine and fecal samples
Metabolite Profiling | approximately 11 days
  To provide plasma, urine and faecal samples for metabolite profiling and structural identification
Total radioactivity in plasma PK:Tmax | approximately 11 days
  Time for Cmax
Total radioactivity in plasma PK:AUC0-t | approximately 11 days
  Area under the plasma concentration time profile from time 0 to time of the last quantifiable concentration.
Total radioactivity in plasma PK:t1/2 | approximately 11 days
  Elimination half-life.
Total radioactivity in plasma PK:CL/F | approximately 11 days
  Drug clearance
Total radioactivity in plasma PK:Vd/F | approximately 11 days
  Apparent volume of distribution following oral administration
LXI-15028 and metabolite PK:Cmax | approximately 11 days
  Maximum plasma concentration
LXI-15028 and metabolite PK:Tmax | approximately 11 days
  Time for Cmax
LXI-15028 and metabolite PK:AUC0-t | approximately 11 days
  Area under the plasma concentration time profile from time 0 to time of the last quantifiable concentration.
LXI-15028 and metabolite PK:AUC0-inf | approximately 11 days
  Area under the plasma concentration time profile from time 0 to infinity.
LXI-15028 and metabolite PK:t1/2 | approximately 11 days
  Elimination half-life.
LXI-15028 and metabolite PK:CL/F | approximately 11 days
  Drug clearance
LXI-15028 and metabolite PK:Vd/F | approximately 11 days
  Apparent volume of distribution following oral administration

SECONDARY OUTCOMES:
Adverse events | approximately 11 days
  Number of adverse events, which are any untoward medical occurrence regardless of attribution to study drug in a participant who received study drug

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miu, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

REFERENCES:
- [Derived] Bian Y, Yuan J, Ma S, Nan J, Gu Z, Feng H, Yu Z, Liu Z, Xie F, Wang Y, Liu C, Zhang H, Miao L. Mass balance and metabolite profiles in humans of tegoprazan, a novel potassium-competitive acid blocker, using 14C-radiolabelled techniques. Expert Opin Drug Metab Toxicol. 2025 Jul;21(7):897-907. doi: 10.1080/17425255.2025.2505637. Epub 2025 May 13. PMID 40349123